CLINICAL TRIAL: NCT05450627
Title: Development of a Registry of Patients With Pancreatic Exocrine Insufficiency of Different Etiologies
Brief Title: Registry of Pancreatic Exocrine Insufficiency.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Responsible Party: Principal Investigator, J. Enrique Domínguez-Muñoz, Head of the Department of Gastroenterology, Hospital Clinico Universitario de Santiago
Other Study IDs: PEI-01-2021
Record Dates: First submitted 2022-07-05; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Exocrine Pancreatic Insufficiency
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Case: Adult patients diagnosed with pancreatic exocrine insufficiency of any etiology
  Interventions: Drug: Pancreatic Enzyme

INTERVENTIONS:
Drug: Pancreatic Enzyme — Registry of pancreatic enzyme therapy prescribed to included patients

SUMMARY:
A prospective, cross-sectional, observational study has been designed with the aim of the study is to evaluate the diagnosis and management of patients with pancreatic exocrine insufficiency secondary to different pancreatic diseases and conditions in clinical practice.

A registry has been develop to include patients older than 18 years diagnosed with pancreatic exocrine insufficiency, sho are willing to participate in the study and sign the informed consent.

Registry includes demographics, toxic habits,pharmacological therapies, underlying disease that causes pancreatic exocrine insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years diagnosed with PEI secondary to pancreatic diseases, pancreatectomy, or gastrectomy.
* Willingness to participate in the study.

Exclusion Criteria:

* Patients with pancreatic diseases without PEI.
* Pregnancy
* Known allergy to oral pancreatic enzymes
* Any condition avoiding adequate clinical management of PEI.
* Patients who are not willing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with pancreatic exocrine insufficiency of any etiology.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose of oral pancreatic enzymes | Six months
  Dose required for symptoms relief and normalization of the nutritional status

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico Universitario de Santiago, Santiago de Compostela, A Coruña, Spain